CLINICAL TRIAL: NCT07407062
Title: Folate Receptor Alpha Expression in Relapsed Ovarian, Fallopian Tube and Primary Peritoneal Cancer: a Realworld prEvalence Study in Italy
Brief Title: A Study to Evaluate Folate Receptor Alpha (FRα) Expression in Adult Participants With Ovarian, Fallopian Tube, and Primary Peritoneal Cancer in Italy
Acronym: FORCE
Status: Not yet recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H26-138
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cancer - Ovarian
Keywords: Cancer - Ovarian
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived surgical tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Folate Receptor Alpha (FRα): Samples of eligible participants with ovarian cancer will be analyzed retrospectively for folate receptor alpha (FRα) expression.

SUMMARY:
The purpose of this study is to evaluate the prevalence of folate receptor alpha (FRα)-positive status (≥75% viable tumor cells with moderate (2+) and/or strong (3+) membrane staining) in participants with high-grade serous ovarian, fallopian tube, and primary peritoneal cancer, stratified by time of sampling (initial diagnosis versus relapse), adhering to Ventana folate receptor alpha (FOLR1) RxDx (prescription diagnosis) assay Interpretation Guidance.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed ovarian, fallopian tube and primary peritoneal cancer
* Histologically high-grade serous carcinoma
* Presence of archived surgical tissue samples from participants with epithelial ovarian cancer at diagnosis and at 1st recurrence in the same participants
* Available samples collected from January 1st, 2016 to study start date (defined as study site initiation visit date) that are considered adequate for the Ventana folate receptor alpha (FOLR1) RxDx assay by the site pathologist

Exclusion Criteria:

* Histological ambiguous diagnosis upon review
* Diagnosis based on cytology and without any biopsy or surgical specimen
* Other histotypes than high grade serous ovarian cancer, fallopian tube cancer and primary peritoneal cancer
* Archival or recurrent sample for the same participant not available

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed on archived tissue samples from approximately 200 eligible female adult participants with relapsed high grade serous epithelial ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
FRα - Positive Status | Up to Approximately 6 Months
  FRα - positive status, defined as ≥75% viable tumor cells demonstrating moderate (2+) and/or strong (3+) membrane staining with the Ventana FOLR1 RxDx assay, at diagnosis and/or at relapse.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=H26-138